CLINICAL TRIAL: NCT01446419
Title: A Prospective Randomized, Double-blind, Controlled Investigation Evaluating the Intracept Intraosseous Nerve Ablation System for the Reduction of Pain in Patients With Chronic Axial Low Back Pain
Brief Title: SMART Clinical Study: Surgical Multi-center Assessment of RF Ablation for the Treatment of Vertebrogenic Back Pain
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Relievant Medsystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CIP 0003
Record Dates: First submitted 2011-10-03; First posted 2011-10-05 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Low Back Pain
Keywords: chronic axial low back pain; vertebrogenic pain; Radio frequency ablation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intracept Treatment (Experimental)
  Interventions: Device: Intracept Treatment
- Sham Treatment (Sham Comparator)
  Interventions: Device: Sham Treatment

INTERVENTIONS:
Device: Intracept Treatment — Percutaneous transpedicular RF ablation of an intraosseous nerve within the lumbar vertebral body to treat chronic axial low back.
  Arms: Intracept Treatment
Device: Sham Treatment — Percutaneous transpedicular access to the lumbar vertebra, no RF ablation delivered.
  Arms: Sham Treatment

SUMMARY:
To evaluate the safety and efficacy of RF ablation using the Intracept Intraosseous Nerve Ablation System to ablate intraosseous nerves for the relief of chronic axial low back pain. This is a prospective, double-blind, randomized, sham-controlled clinical trial with an optional crossover component.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature patients age 25 - 70 years, inclusive
* Chronic lower back pain for at least six (6) months
* Failure to respond to at least six (6) months of non-operative conservative management. The minimum requirement is as follows:

  * Analgesic therapy (minimum of 2 weeks) and a minimum of 4 weeks of NSAID therapy
  * Supervised exercise program(minimum of 12 sessions)
* Oswestry Disability Index (ODI) at time of evaluation of at least 30 points
* Baseline Visual Analog Scale (VAS) of at least 4cm on a 10cm scale
* The following test indicating that the vertebral body is the source of pain:

  1.MRI showing Type 1 or Type II Modic changes at least one vertebral endplate, at one or more levels from L3 to S1
* Understands the local language and is willing and able to follow the requirements of the protocol
* Understands the informed consent and signs the institutional review board/ independent ethics committee (IRB/IEC) approved informed consent form

Exclusion Criteria:

* Radicular pain by history or evidence of pain or neurological deficit in a dermatomal zone at or below the medial thigh.
* Previous surgery performed on the lumbar spine
* History of symptomatic spinal stenosis
* History of osteoporotic or tumor-related vertebral body compression fracture
* History of vertebral cancer or spinal metastasis
* History of spinal infection
* Metabolic bone disease (e.g. osteogenesis imperfecta)
* BMI ≥40
* Osteoporosis, defined as T score <-2.5
* Any radiographic evidence of other important back pathology, such as:

  1. Nerve root compression or severe effacement of the thecal sac that correlates with radicular pain or muscle weakness
  2. Disc extrusion or disc protrusion >5mm
  3. Facet arthrosis or facet effusion at any lumbar level that correlates with clinical evidence of facet mediated low back pain
  4. Spondylolisthesis 2mm or greater at any level
  5. Spondylolysis at any level
* MRI evidence of Modic changes, Type I or Type II at greater than 3 vertebral bodies.
* Any back pathology related to trauma, evidence of vertebral compression fracture or other spinal pathology that could affect assessment of response to back pain
* Demonstrates 3 or more Waddell's signs of Inorganic Behavior
* Any evidence of current systemic infection
* Uncorrected bleeding diathesis
* Any neurologic problem that prevents early mobilization after surgery or interferes with assessment of ODI
* Contraindication to MRI or patients who have allergies to the components of the Intracept device
* Pregnant, lactating or plan to become pregnant in next year
* Diabetes requiring daily insulin
* Current use of steroid therapy, with the exception of inhalation steroids for asthma
* Evidence of mental instability or uncontrolled depression; patients requiring anti-depressants or anti-psychotics within 3 months of enrollment are not eligible; patients with a Beck Depression Score of greater than 24 are not eligible
* Receiving Workmen's Compensation
* Currently involved in litigation regarding back pain/injury or financial incentive to remain impaired
* Any medical condition that impairs follow-up
* Contraindications to the proposed anesthetic protocol.
* Evidence of substance abuse; patients using prescribed extended release narcotics are not eligible (e.g. fentanyl patch,MS contin, oxycontin)
* Known to require at the time of screening and/or randomization, additional surgery to the lumbar spinal region within six months
* Being treated with radiation, chemotherapy, immunosuppression, or chronic steroid therapy (prednisone use up to 5 mg/qd or its equivalent is allowed)
* Has a life expectancy of less than 1 year
* Has active implantable devices, such as cardiac pacemakers, spinal cord stimulators, etc.
* Is a prisoner

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2011-10; Primary Completion 2015-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Fischgrund, MD, Principal Investigator — Michigan Orthopaedic Institute
Locations (13):
- United States (13):
  - Desert Institute for Spine Care, Phoenix, Arizona
  - SpineCare Medical Group, Daly City, California
  - Memorial Orthopedic Surgical Group, Long Beach, California
  - The Spine Institute, Santa Monica, California
  - Pain Center Solutions, Marietta, Georgia
  - Indiana Spine Group, Carmel, Indiana
  - Maine Medical Partners, Scarborough, Maine
  - Partners in Research and Educational Studies of Spinal Disorders (PressD), Southfield, Michigan
  - OrthoCarolina, Charlotte, North Carolina
  - NeuroSpine Institute, Eugene, Oregon
  - Rothman Institute, Philadelphia, Pennsylvania
  - Seton Spine & Scoliosis Center, Austin, Texas
  - Virginia iSpine Physicians, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at 15 sites in the US and 3 sites in Germany
Pre-assignment Details: 2:1 Randomization (treatment: sham)
Groups:
- Intracept Treatment: Intracept Treatment: Percutaneous access and RF ablation of the basivertebral nerve within the lumbar vertebral body to treat chronic axial low back.
- Sham Treatment: Sham Treatment: Percutaneous access to the lumbar vertebra, no RF ablation delivered.
Period: Overall Study
Arm/Group | Intracept Treatment | Sham Treatment
Started | 147 | 78
3 Month Follow-up | 146 | 77
6 Month Follow-up | 144 | 77
12 Month Follow-up | 142 | 77
Completed | 142 | 77
Not Completed | 5 | 1
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Terminated per protocol | 3 | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Intracept Treatment | Sham Treatment | Total
Number analyzed (Participants) | 147 | 78 | 225
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 138 | 74 | 212
  >=65 years | 9 | 4 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (10.46) | 47.1 (8.97) | 47.0 (9.95)
Gender [Count of Participants; unit: Participants]
  Female | 65 | 37 | 102
  Male | 82 | 41 | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 5 | 14
  Not Hispanic or Latino | 138 | 73 | 211
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 134 | 71 | 205
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 133 | 69 | 202
  Germany | 14 | 9 | 23
Oswestry Disability Index (ODI) [Mean (Standard Deviation); unit: units on a scale] — ODI is a patient questionnaire that assesses back dysfunction due to back pain. There are 10 questions that are scored from 0-5. The obtained score is multiplied by 2 to produce a percentage score that is reported on a scale of 0-100. Scores are interpreted as follows: 0-20% minimum disability; 21-40% moderate disability; 41-60% severe disability; 61-80% crippled; 81-100% bed bound or exaggerating their symptoms.
  units on a scale | 42.9 (10.73) | 41.1 (10.39) | 42.2 (10.63)

OUTCOME MEASURES:

1. Primary Outcome: Change in ODI From Baseline to 3 Months Post-treatment
Description: The primary variable is the Oswestry Disability Index (ODI) and the primary efficacy endpoint is the mean improvement from baseline to 3 months in the ODI. The primary endpoint will be evaluated in both the treatment and sham groups with between-group comparisons used to assess the success of the Intracept System in reducing chronic axial low back pain.
  ODI is a patient questionnaire that assesses back dysfunction due to back pain. There are 10 questions that are scored from 0-5. The obtained score is multiplied by 2 to produce a percentage score that is reported on a scale of 0-100. Scores are interpreted as follows: 0-20% minimum disability; 21-40% moderate disability; 41-60% severe disability; 61-80% crippled; 81-100% bed bound or exaggerating their symptoms.
Time Frame: 3 months
Population: Per Protocol Population: subjects that received the intended therapy per randomization assignment (appropriate ablation of the basivertebral nerve in the Intracept System arm) and completed follow-up per the study protocol.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intracept Treatment | Sham Treatment
Number analyzed (Participants) | 128 | 77
units on a scale | -20.5 [-23.2 to -17.8] | -15.2 [-18.7 to -11.7]
Statistical Analysis 1: Comparison: Intracept Treatment vs Sham Treatment; Test type: Superiority or Other; p = 0.019, ANCOVA; P-value from ANCOVA with factors of tx group, analysis center and tx group by analysis center interaction, and a covariate of baseline ODI score

2. Secondary Outcome: Patient Success at 3 Months
Description: Proportion of subjects with clinical success at 3 months, where clinical success was defined as:
  * 3 month ODI score represented at least a 15-point reduction from baseline
  * no device or procedure related SAE between baseline and 3 mos.
  * no increase in opioid use between procedure and 3 mos.
  * no deficit in a motor or dermatomal sensory group at the treated level at 3 mos.
  * no operative interventions or invasive procedures for lumbar back pain by a pain management or spinal specialist between procedure and 3 mos.
Time Frame: 3 months
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Intracept Treatment | Sham Treatment
Number analyzed (Participants) | 128 | 77
percentage of patients | 55.5 | 45.5

3. Secondary Outcome: Change in ODI From Baseline to 6 Months Post-treatment
Description: The improvement in ODI at 6 months compared to baseline.
  ODI is a patient questionnaire that assesses back dysfunction due to back pain. There are 10 questions that are scored from 0-5. The obtained score is multiplied by 2 to produce a percentage score that is reported on a scale of 0-100. Scores are interpreted as follows: 0-20% minimum disability; 21-40% moderate disability; 41-60% severe disability; 61-80% crippled; 81-100% bed bound or exaggerating their symptoms.
Time Frame: 6 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intracept Treatment | Sham Treatment
Number analyzed (Participants) | 128 | 77
units on a scale | -20.8 [-23.4 to -18.2] | -17.0 [-20.3 to -13.7]

ADVERSE EVENTS:
Time Frame: 12 Months
Description: Adverse Events reported for all Intent to Treat subjects from randomization through 12 months of follow-up
Arm/Group | Intracept Treatment | Sham Treatment
Serious Adverse Events (participants affected / at risk) | 9/147 | 5/78
Other Adverse Events (participants affected / at risk) | 78/147 | 24/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intracept Treatment (N=147) | Sham Treatment (N=78)
Gastrointestinal bacterial infection (Infections and infestations) | 1 (1) | 0 (0) — Not related to device or procedure
Airway obstruction on anaesthetic induction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Procedure related
Complications from lymph node excision (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Not related to device or procedure
Arthritis aggravated (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Not related to device or procedure
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Not related to device or procedure
Low back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — Not related to device or procedure
Grand mal seizure (Nervous system disorders) | 1 (1) | 0 (0) — Not related to device or procedure
CVA (Nervous system disorders) | 0 (0) | 1 (1) — Not related to device or procedure
C-section (Surgical and medical procedures) | 0 (0) | 1 (1) — Not related to device or procedure
Hip replacement (Surgical and medical procedures) | 1 (1) | 1 (1) — Not related to device or procedure
Bladder operation (Surgical and medical procedures) | 1 (1) | 0 (0) — Not related to device or procedure
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) — Not related to device or procedure
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intracept Treatment (N=147) | Sham Treatment (N=78)
Incision site discomfort (Injury, poisoning and procedural complications) | 17 (17) | 5 (5)
Leg pain (Musculoskeletal and connective tissue disorders) | 12 (12) | 4 (4)
Low back pain (Musculoskeletal and connective tissue disorders) | 34 (35) | 11 (11)
Post procedural nausea (Injury, poisoning and procedural complications) | 15 (15) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Individual PIs will not publish any study results until completion of study and publication of the multi-center results in a peer-reviewed journal, which shall occur within one year after study completion. Thereafter, PIs may publish individual site experience. Sponsor can review results communications prior to public release and can embargo communications regarding results for a period that is less than or equal to 60 days from the time submitted to sponsor for review.